CLINICAL TRIAL: NCT04518306
Title: Efficacy and Safety of GMRx2 (a Single Pill Combination Containing Telmisartan/Amlodipine/Indapamide) Compared to Placebo for the Treatment of Hypertension
Brief Title: Efficacy and Safety of GMRx2 Compared to Placebo for the Treatment of Hypertension
Acronym: GMRx2_PCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: George Medicines PTY Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMRx2-HTN-2020-PCT1
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine; Indapamide

STUDY DESIGN:
Intervention Model Description: International, multicenter, randomized, double-blind, placebo-controlled, parallel-group trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Triple ¼ (GMRx2) (Experimental): Telmisartan 10 mg/amlodipine 1.25 mg/indapamide 0.625 mg
  Interventions: Drug: Telmisartan 10 mg/amlodipine 1.25 mg/indapamide 0.625 mg
- Triple ½ (GMRx2) (Active Comparator): Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg
  Interventions: Drug: Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan 10 mg/amlodipine 1.25 mg/indapamide 0.625 mg — Oral tablets
  Arms: Triple ¼ (GMRx2)
Drug: Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg — Oral tablets
  Arms: Triple ½ (GMRx2)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Recent hypertension guidelines recommend combination therapy as initial treatment for many or most patients. Several trials suggest triple low-dose combination therapy may be highly effective in terms of achieving blood pressure control without increasing adverse effects. This trial is designed to investigate the efficacy and safety of GMRx2 in participants with high blood pressure compared to placebo.

DETAILED DESCRIPTION:
TRIAL DRUG:

GMRx2: single pill combination of telmisartan/amlodipine/indapamide Dose version 1: telmisartan 10 mg/amlodipine 1.25 mg/indapamide 0.625 mg Dose version 2: telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg INDICATION: Hypertension

TRIAL TITLE:

Efficacy and safety of GMRx2 compared to placebo for the treatment of hypertension.

OBJECTIVES:

To investigate the efficacy and safety of GMRx2 compared to placebo for the treatment of hypertension.

INTERVENTION:

A 2-week single-blind placebo run-in will be followed by a 4-week double-blind period with randomization to GMRx2 dose version 1, GMRx2 dose version 2 or placebo.

ELIGIBILITY:
Inclusion Criteria

At screening visit:

1. Provided signed consent to participate in the trial.
2. Adult aged ≥18 years.
3. Low calculated CV risk according to local guidelines such that pharmacological BP-lowering treatment is not mandatory: e.g. Pooled Cohorts Equation 10-years ASCVD risk <10% in the USA.
4. Likely diagnosis of hypertension, defined as one or more of:

   * automated SBP at this clinic visit according to trial methods (see Appendix 2) of ≥130mmHg on no BP lowering medicines or ≥120mmHg on 1 BP lowering medicine that will be stopped at this visit, OR
   * documentation in last 6 months of office SBP ≥ 140 mmHg and/or DBP ≥ 90mmHg on no BP lowering medicines or SBP ≥ 130 mmHg and/or DBP ≥ 85mmHg on 1 BP lowering medicine that will be stopped at this visit, OR
   * documentation in last 6 months of home SBP ≥ 130 mmHg and/or DBP ≥ 80mmHg on no BP lowering medicines or SBP ≥ 120 mmHg and/or DBP ≥ 75mmHg on 1 BP lowering medicine that will be stopped at this visit, OR
   * documentation in last 6 months of ambulatory daytime SBP ≥ 130 mmHg and/or DBP ≥ 80mmHg on no BP lowering medicines or SBP ≥ 120 mmHg and/or DBP ≥ 75mmHg on 1 BP lowering medicine that will be stopped at this visit
5. No contraindication to trial medications, including 2-weeks placebo run-in and 4-weeks randomized treatment period with GMRx2 (dose version 1 or 2) or placebo.

At randomization visit:

1. Home seated mean SBP 130-154 mmHg in the week before the randomization visit.
2. Adherence of 80-120% to placebo run-in.
3. Tolerated placebo run-in.
4. Adherence to home BP monitoring schedule: in the week before randomization, at least 6 measures (e.g. ≥2 sets of triplicate measures) including at least 1 morning and 1 evening each with ≥2 measures. Morning is defined as any measure in the am and evening as any measure in the pm. Morning and evening do not have to be same day.

Exclusion Criteria:

At screening visit:

1. Receiving 2 or more BP-lowering drugs.
2. Clinic seated mean SBP ≥160 mmHg and/or DBP ≥100 mmHg.
3. Pregnant or had a positive pregnancy test or unwilling to undertake a pregnancy test during the trial and up to 30 days after the discontinuation of the trial medication or breastfeeding or of childbearing age and not using an acceptable method of contraception. Acceptable methods of birth control include hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (e.g. condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization. Contraception should be used for at least 1 month before the screening visit and until the end of trial participation.
4. Not suitable for participation in a clinical trial according to local ethical or regulatory requirements related to severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2).
5. Contraindication, including hypersensitivity (e.g. anaphylaxis or angioedema), to any of the 3 trial medications.
6. Current/history of transient ischemic attack, stroke, or hypertensive encephalopathy.
7. Current/history of acute coronary syndrome, unstable angina, myocardial infarction, percutaneous transluminal coronary revascularization, or coronary artery bypass graft.
8. Current/history of New York Heart Association class III and IV congestive heart failure.
9. Current/history of a known secondary cause of hypertension, such as primary aldosteronism, renal artery stenosis, pheochromocytoma, or Cushing's syndrome.
10. Current/history of substantially uncontrolled diabetes (HbA1c > 11.0%) within last three months.
11. Current/history of end-stage renal disease or anuria or estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2.
12. Current/history of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the upper limit of normal range within 6 months.
13. Current concomitant illness or physical impairment or mental condition that in the judgment of the investigator could interfere with the effective conduct of the trial or constitutes a significant risk to the participants' well-being.
14. Arm circumference that is too large (>55 cm) or too small (<20 cm) to allow accurate measurement of BP.
15. Currently taking or might need during the trial, a concomitant treatment which is known to interact significantly with the trial medication: digoxin, lithium, diabetics receiving aliskiren, moderate and strong CYP3A4 inhibitors [e.g. ritonavir, ketoconazole, diltiazem], simvastatin >20 mg/day, immunosuppressants.
16. Might need treatment with drugs that are prohibited during the trial: other antihypertensive drugs, endothelin receptor antagonists, neprilysin inhibitors, or other drugs that may affect BP (see Error! Reference source not found.).
17. Current surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of trial drugs such as prior major gastrointestinal tract surgery (e.g. gastrectomy, lap band, or bowel resection) or acute flare of inflammatory bowel disease within one year.
18. Individuals working >2-night shifts per week.
19. Participated in any investigational drug or device trial within the previous 30 days.
20. History of alcohol or drug abuse within 12 months.

At randomization visit:

1. Unable to adhere to the trial procedures during the run-in period.
2. Any of the following which in the investigator's judgment may compromise the safety of the participant if randomized to the trial medications:

   1. High or low clinic BP levels even in the light of the values for home BP that are available for that participant. The exact levels of BP are not specified, since there is clinical uncertainty as to the relevance of BP levels which are high/low in clinic only; for example the clinical relevance of 'whitecoat hypertension' is uncertain.
   2. High or low home DBP levels. The exact levels of DBP are not specified, reflecting clinical uncertainty of for example isolated diastolic hypertension. However, home DBP values of >99 mmHg may typically be considered as requiring treatment intensification, and such participants would not be suitable for randomization.
3. Any abnormal laboratory value which in the judgment of the investigator could interfere with the effective conduct of the trial or constitutes a significant risk to the participants' well-being.
4. Fulfilling any of the exclusion criteria mentioned for the screening visit, when verified again at randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Rodgers, Professor, Principal Investigator — The George Institute
Locations (46):
- United States (22):
  - Elite Clinical Studies, Phoenix, Arizona
  - Headlands Research, Scottsdale, Arizona
  - Quality of Life Medical & Research Centers, LLC, Tucson, Arizona
  - Valiance Clinical Research, South Gate, California
  - Valiance Clinical Research, Tarzana, California
  - Clinical Research of Brandon, Brandon, Florida
  - Inpatient Research Clinic, Hialeah, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Ocala Research Institute, Ocala, Florida
  - Altus Research, Inc, Palm Beach, Florida
  - Suncoast Research Associates, St. Petersburg, Florida
  - Accel Research, St. Petersburg, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Precision Research Center, Tampa, Florida
  - Buckhead Primary Care Research, Snellville, Georgia
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - Synergy Groups Medical, Houston, Texas
  - Synergy Groups Medical, Missouri City, Texas
  - North Hills Medical Research, North Richland Hills, Texas
  - Meridian Clinical Research, Portsmouth, Virginia
- Australia (5):
  - Castle Hill Medical Centre, Castle Hill, New South Wales
  - Hudson Institute of Medical Research, Clayton, Victoria
  - Barwon Health, Geelong University Hospital, Geelong, Victoria
  - Curtin University, Bentley, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Nigeria (2):
  - University of Abuja Teaching Hospital, Gwagwalada, Federal Capital Territory
  - Aminu Kano Teaching Hospital, Kano
- Sri Lanka (7):
  - Institute of Cardiology, National Hospital of Sri Lanka, Colombo
  - Colombo South Teaching Hospital, Dehiwala
  - Karapitiya Teaching Hospital, Galle
  - Jafna Teaching Hospital, Jaffna
  - Kandy National Hospital, Kandy
  - Kurunegala Teaching Hospital, Kurunegala
  - Colombo North Teaching Hospital, Ragama
- United Kingdom (10):
  - Steploe Medical Centre, Soham, Cambridgeshire
  - Newquay Medical, Newquay, Cornwall
  - Burbage Surgery, Hinckley, Leicestershire
  - Belmont Health Centre, Harrow, London
  - West Walk Surgery, Bristol, Somerset
  - Brockwood Medical Practice, Betchworth, Surrey
  - Lakeside Surgery, Coventry, West Midlands
  - Trowbridge Health Centre, Trowbridge, Wiltshire
  - Abbeywell Surgery, Romsey
  - Albany House Medical Centre, Wellingborough

IPD SHARING:
Plan to Share IPD: No
No If the sponsor receives a request for study data, then such requests will be reviewed by sponsor following completion of regulatory submissions and review, and with support from members of the GMRX2 steering committee who will advise on the scientific merit and integrity of the proposed analysis.

REFERENCES:
- [Derived] Salam A, de Silva HA, Ojji D, de Silva AP, Galappatthy G, Lakshman P, Kumanan T, Mayurathan G, Pereira T, Rahuman M, Ranasinghe G, Rasnayake L, Uluwattage W, Constantine GR, Kandeepan T, Sani MU, Kumar A, Pant R, Cushman WC, Di Tanna GL, Grobbee D, Narkiewicz K, Oparil S, Poulter NR, Schlaich MP, Schutte AE, Spiering W, Williams B, Wright JT Jr, Gianacas C, Shanthakumar M, Liu X, Freed R, Whelton PK, Rodgers A. Long-Term Efficacy and Safety of a Novel Low-Dose Triple Single-Pill Combination for the Treatment of Hypertension. Glob Heart. 2025 Oct 31;20(1):102. doi: 10.5334/gh.1481. eCollection 2025. PMID 41180852
- [Derived] Rodgers A, Salam A, Schutte AE, Cushman WC, de Silva HA, Di Tanna GL, Grobbee D, Narkiewicz K, Ojji DB, Poulter NR, Schlaich MP, Oparil S, Spiering W, Williams B, Wright JT Jr, Gutierez A, Sanni A, Lakshman P, McMullen D, Ranasinghe G, Gianacas C, Shanthakumar M, Liu X, Wang N, Whelton P. Efficacy and Safety of a Novel Low-Dose Triple Single-Pill Combination Compared With Placebo for Initial Treatment of Hypertension. J Am Coll Cardiol. 2024 Dec 10;84(24):2393-2403. doi: 10.1016/j.jacc.2024.08.025. Epub 2024 Aug 31. PMID 39217570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 47 trial centers spread across 5 countries (United States of America [USA] 23, Great Britain 10, Sri Lanka 7, Australia 5, and Nigeria 2).
Pre-assignment Details: Out of 1584 participants screened, 755 participants entered the 2-week single-blind placebo run-in period. Overall, 460 of the 755 participants who entered the run-in period were not randomized, the most common reason was failure to meet the criteria of home seated mean SBP of 130-154 mmHg in the week prior to the randomization visit. Total of 295 participants were randomized to the treatment groups at the end of run-in period.
Groups:
- Triple ¼ (GMRx2): Telmisartan 10 mg/amlodipine 1.25 mg/indapamide 0.625 mg
  Telmisartan 10 mg/amlodipine 1.25 mg/indapamide 0.625 mg: Oral tablets
  Over encapsulated Telmisartan 10 mg/amlodipine 1.25 mg/indapamide 0.625 mg oral tablet once daily in the morning after home blood pressure (BP) measurement from week 1 to week 4
- Triple ½ (GMRx2): Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg
  Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg: Oral tablets
  Over encapsulated Telmisartan 20 mg/amlodipine 2.5 mg/indapamide 1.25 mg oral tablet once daily in the morning after home BP measurement from week 1 to week 4
- Placebo: Placebo
  Placebo: Placebo
  One tablet daily in the morning after home BP measurement from week 1 to week 4.
Period: Single-Blind Placebo Run-In Period
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Started | 0 | 0 | 755
Completed (Enrolled participants completed single-blind run-in period on placebo and were subsequently randomized to blinded treatment arms.) | 0 | 0 | 295
Not Completed | 0 | 0 | 460
Period: Double-Blind Period
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Started | 113 | 119 | 63
Completed | 91 | 91 | 50
Not Completed | 22 | 28 | 13
Not completed — Run in failure | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Participant moved to open-label extension (OLE) study | 21 | 21 | 8
Not completed — Other | 0 | 2 | 0
Not completed — Missing | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized on the safety population by randomized treatment groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo | Total
Number analyzed (Participants) | 113 | 119 | 63 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.25) | 51.2 (9.88) | 50.9 (12.81) | 50.5 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 61 | 36 | 165
  Male | 45 | 58 | 27 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 42 | 23 | 105
  Not Hispanic or Latino | 70 | 76 | 38 | 184
  Unknown or Not Reported | 3 | 1 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 26 | 27 | 8 | 61
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 18 | 20 | 11 | 49
  White | 66 | 72 | 43 | 181
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59 | 65 | 33 | 157
  Sri Lanka | 19 | 18 | 6 | 43
  United Kingdom | 18 | 15 | 10 | 43
  Australia | 15 | 16 | 11 | 42
  Nigeria | 2 | 5 | 3 | 10
Height [Mean (Standard Deviation); unit: cm] | 165.97 (10.439) | 166.68 (10.247) | 167.36 (9.878) | 166.55 (10.223)
Weight [Mean (Standard Deviation); unit: kg] | 85.50 (20.865) | 85.12 (22.419) | 84.92 (20.299) | 85.22 (21.319)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (6.04) | 30.4 (6.69) | 30.0 (5.67) | 30.5 (6.22)
Smoking - Never [Count of Participants; unit: Participants] | 90 | 79 | 47 | 216
Smoking - Ex-smoker [Count of Participants; unit: Participants] | 15 | 28 | 12 | 55
Smoking - Current smoker [Count of Participants; unit: Participants] | 8 | 12 | 4 | 24
Alcohol consumption - Currently drink alcohol once a week or more [Count of Participants; unit: Participants] | 38 | 50 | 25 | 113
Pre-screening 12-lead ECG - Normal [Count of Participants; unit: Participants] | 83 | 87 | 47 | 217
Pre-screening 12-lead ECG - Any other abnormalities [Count of Participants; unit: Participants] | 30 | 32 | 16 | 78
Education - No formal education [Count of Participants; unit: Participants] | 0 | 0 | 1 | 1
Education - Primary school [Count of Participants; unit: Participants] | 7 | 8 | 5 | 20
Education - Secondary school [Count of Participants; unit: Participants] | 33 | 39 | 13 | 85
Education - Tertiary school [Count of Participants; unit: Participants] | 52 | 57 | 39 | 148
Vocational training [Count of Participants; unit: Participants] | 21 | 15 | 5 | 41

OUTCOME MEASURES:

1. Primary Outcome: Difference in Change in Home Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 4
Description: Each blood pressure (BP) measurement consisted of valid SBP values (ie. SBP>60 mmHg and <250 mmHg). BP values were summarized using descriptive statistics, including actual values and changes from randomization to Week 4, by timepoint and treatment groups.
Time Frame: Randomization to Week 4
Population: Analysis was performed on randomized set (All participants who have been randomized). Participants were analyzed in the treatment group to which they have been randomized.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
mmHg | -9.6 (1.00) | -10.4 (1.33) | -2.2 (1.16)
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; The analysis was performed using a mixed model for repeated measures (MMRM) for estimating the difference between Triple ¼ GMRx2 and placebo at Week 4; Test type: Superiority; p < 0.0001, MIANALYZE procedure — No adjustment for multiplicity was made and the 0.05 level of significance was used to claim efficacy compared with placebo; LS Means Difference = -7.33, 95% CI 2-sided [-10.176 to -4.486], Standard Error of Mean 1.451
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; The analysis was performed using a mixed model for repeated measures (MMRM) for estimating the difference between Triple ½ GMRx2 and placebo at Week 4; Test type: Superiority; p < 0.0001, MIANALYZE procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -8.23, 95% CI 2-sided [-11.305 to -5.151], Standard Error of Mean 1.570

2. Secondary Outcome: Difference in Change in Clinic Seated Mean Mean Systolic Blood Pressure (SBP) From Randomization to Week 4
Description: as for outcome 1
Time Frame: Randomization to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
mmHg | -6.6 (0.94) | -8.2 (1.25) | 1.3 (1.19)
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -7.98, 95% CI 2-sided [-11.281 to -4.681], Standard Error of Mean 1.649
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -9.52, 95% CI 2-sided [-13.588 to 5.449], Standard Error of Mean 2.034

3. Secondary Outcome: Difference in Change in Clinic Seated Mean Diastolic Blood Pressure (DBP) From Randomization to Week 4
Description: Each blood pressure (BP) measurement consisted of valid DBP values (ie. DBP>40mmHg and <150mmHg). BP values were summarized using descriptive statistics, including actual values and changes from randomization to Week 4, by timepoint and treatment groups.
Time Frame: Randomization to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
mmHg | -3.5 (0.60) | -4.3 (0.93) | 0.5 (0.91)
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; p = 0.0015, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -4.00, 95% CI 2-sided [-6.413 to -1.597], Standard Error of Mean 1.204
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -4.86, 95% CI 2-sided [-7.130 to -2.595], Standard Error of Mean 1.133

4. Secondary Outcome: Percentage of Participants With Clinic Seated Mean Systolic Blood Pressure (SBP) <140 and DBP <90 mmHg at Week 4
Description: The percentage of participants achieving averaged clinic SBP <140 and DBP <90 mmHg at Week 4 was evaluated.
Time Frame: At Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 73 | 83 | 23
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; p = 0.0002, Wald test; Risk Difference (RD) = 28.09, 95% CI 2-sided [11.811 to 42.450] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, Wald test; Risk Difference (RD) = 33.24, 95% CI 2-sided [17.199 to 47.186] — 95% confidence intervals for risk difference utilize Newcombe estimation method

5. Secondary Outcome: Percentage of Participants With Clinic Seated Mean Systolic Blood Pressure (SBP) <130 and Diastolic Blood Pressure (DBP) <80 mmHg at Week 4
Description: The percentage of participants achieving averaged clinic SBP <130 and DBP <80 mmHg at Week 4 was evaluated. Participants were analyzed in the treatment group to which they have been randomized.
Time Frame: At Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 23 | 36 | 2
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Percentages were calculated from the total number of participants within the randomized set; Test type: Superiority; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 17.18, 95% CI 2-sided [6.070 to 26.385] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Percentages were calculated from the total number of participants within the randomized set; Test type: Superiority; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 27.08, 95% CI 2-sided [15.237 to 36.646] — 95% confidence intervals for risk difference utilized Newcombe estimation method

6. Secondary Outcome: Difference in Change in Home Seated Mean Diastolic Blood Pressure (DBP) From Randomization to Week 4
Description: Each blood pressure (BP) measurement consisted of valid DBP values (ie. DBP>40mmHg and <150mmHg). BP values were summarized using descriptive statistics, including actual values and changes from randomization to Week 4, by timepoint and treatment groups. To evaluate the difference in change, least squares mean change value is reported.
Time Frame: Randomization to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
mmHg | -5.1 (0.76) | -6.6 (0.60) | -1.1 (0.79)
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; p = 0.0002, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -4.00, 95% CI 2-sided [-5.978 to -2.013], Standard Error of Mean 0.991
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -5.51, 95% CI 2-sided [-7.328 to -3.694], Standard Error of Mean 0.908

7. Secondary Outcome: Difference in Change in Trough Home Seated Mean Systolic Blood Pressure (SBP) From Randomization to Week 4
Description: Difference in change in trough home SBP for GMRx2 vs placebo was evaluated at Week 4. Trough values were measured before morning dose of the study medication.
Time Frame: Randomization to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
mmHg | -8.1 (1.24) | -10.1 (1.36) | -1.3 (1.24)
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; The difference between Triple ¼ GMRx2 Dose and placebo at Week 4 was estimated using MMRM; Test type: Superiority; p = 0.0003, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -6.79, 95% CI 2-sided [-10.300 to -3.287], Standard Error of Mean 1.752
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; The difference between Triple ½ GMRx2 Dose and placebo at Week 4 was estimated using MMRM; Test type: Superiority; p < 0.0001, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -8.74, 95% CI 2-sided [-12.403 to -5.082], Standard Error of Mean 1.829

8. Secondary Outcome: Difference in Change in Trough Home Seated Mean Diastolic Blood Pressure (DBP) From Randomization to Week 4
Description: Difference in change in trough home DBP for GMRx2 vs placebo was evaluated at Week 4. Trough values were measured before morning dose of the study medication. To evaluate the difference in change, least squares mean change value is reported.
Time Frame: Randomization to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
mmHg | -4.2 (0.83) | -5.7 (0.65) | -0.3 (0.93)
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; The difference between Triple ¼ GMRx2 Dose and placebo at Week 4 was estimated using MMRM; Test type: Superiority; p = 0.0003, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -3.86, 95% CI 2-sided [-5.865 to -1.847], Standard Error of Mean 1.004
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; The difference between Triple ½ GMRx2 Dose and placebo at Week 4 was estimated using MMRM; Test type: Superiority; p < 0.0001, MMRM procedure — [p-value comment as in outcome 1, analysis 1]; LS Means Difference = -5.42, 95% CI 2-sided [-7.915 to -2.932], Standard Error of Mean 1.245

9. Secondary Outcome: Percentage of Participants With Home Seated Mean Systolic Blood Pressure (SBP) <135 and Diastolic Blood Pressure (DBP) <85 mmHg at Week 4
Description: The percentage of participants achieving home seated mean SBP <135 and DBP <85 mmHg at Week 4 was evaluated
Time Frame: At Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 67 | 64 | 15
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 35.48, 95% CI 2-sided [19.541 to 48.549] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 29.97, 95% CI 2-sided [14.218 to 43.093] — 95% confidence intervals for risk difference utilized Newcombe estimation method

10. Secondary Outcome: Percentage of Participants With Home Seated Mean Systolic Blood Pressure (SBP) <130 and Diastolic Blood Pressure (DBP) <80 mmHg at Week 4
Description: The percentage of participants achieving averaged home seated mean SBP <130 and DBP <80 mmHg at Week 4 was evaluated
Time Frame: Randomization to Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 32 | 40 | 7
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; p = 0.0030, Wald test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 17.21, 95% CI 2-sided [3.637 to 28.424] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 22.50, 95% CI 2-sided [8.720 to 33.665] — 95% confidence intervals for risk difference utilized Newcombe estimation method

11. Other Pre Specified Outcome: Percentage of Participants Discontinued Trial Medication Due to Adverse Event (AE) or a Serious Adverse Event (SAE) From Randomization to Week 4
Description: The primary safety outcome is percentage of participants discontinued trial medication due to an Adverse Event (AE) or a Serious Adverse Event (SAE) from randomization to Week 4.
Time Frame: Randomization to Week 4
Population: Analysis was done on safety population. The Safety Set is defined as all participants who took at least one dose of study treatment, including during Period 1 single-blind run-in. For the analysis of the safety endpoints, participants were analyzed in the treatment group they actually received. One participant each from Triple ½ (GMRx2) and Placebo group did not receive randomly assigned treatment during "Randomization to Week 4" period.
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 118 | 62
Participants | 0 | 6 | 1
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = -1.61, 95% CI 2-sided [-9.830 to 2.760] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 3.47, 95% CI 2-sided [-5.276 to 9.774] — 95% confidence intervals for risk difference utilized Newcombe estimation method

12. Other Pre Specified Outcome: Percentage of Participants With an Serious Adverse Event (SAE) From Randomization to Week 4
Description: The secondary outcome is percentage of participants with an SAE from randomization to Week 4
Time Frame: Randomization to Week 4
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 118 | 62
Participants | 0 | 2 | 2
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = -3.23, 95% CI 2-sided [-12.171 to 1.662] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = -1.53, 95% CI 2-sided [-10.585 to 4.049]

13. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Hypotension From Randomization to Week 4
Description: The Secondary Safety Outcome is percentage of participants with symptomatic hypotension from randomization to Week 4
Time Frame: Randomization to Week 4
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 118 | 62
Participants | 4 | 6 | 0
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 3.54, 95% CI 2-sided [-4.115 to 9.352] — 95% confidence intervals for risk difference utilize Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 5.08, 95% CI 2-sided [-2.779 to 11.200]

14. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium Concentration Below 135 mmol/l at Week 4
Description: The Secondary safety outcome is percentage of participants with serum sodium concentration below 135 mmol/l at Week 4
Time Frame: At Week 4
Population: The analysis of binary secondary safety endpoints was performed on the Safety Analysis Set, limited to those participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 4 | 1 | 0
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 3.54, 95% CI 2-sided [-4.012 to 9.350] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 0.84, 95% CI 2-sided [-6.364 to 5.278] — 95% confidence intervals for risk difference utilized Newcombe estimation method

15. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium Concentration Above 145 mmol/l at Week 4
Description: The Secondary safety outcome is percentage of participants with serum sodium concentration above 145 mmol/l at Week 4
Time Frame: At Week 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 4 | 5 | 3
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = -1.22, 95% CI 2-sided [-10.928 to 5.573] — 95% confidence intervals for risk difference utilize Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 4.27, 95% CI 2-sided [1.38 to 9.53] — 95% confidence intervals for risk difference utilize Newcombe estimation method

16. Other Pre Specified Outcome: The Percentage of Participants With Serum Potassium Concentration Below 3.5 mmol/l at Week 4
Description: The secondary safety outcome is percentage of participants with serum potassium concentration below 3.5 mmol/l at Week 4
Time Frame: At Week 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 4 | 6 | 1
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 1.95, 95% CI 2-sided [-6.492 to 7.954] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 3.45, 95% CI 2-sided [-5.171 to 9.704] — 95% confidence intervals for risk difference utilized Newcombe estimation method

17. Other Pre Specified Outcome: Percentage of Participants With Serum Potassium Concentration Above 5.5 mmol/l at Week 4
Description: The secondary safety outcome is percentage of participants with serum potassium concentration above 5.5 mmol/l at Week 4.
Time Frame: At Week 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 1 | 0 | 0
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2); Test type: Superiority; Risk Difference (RD) = 0.88, 95% CI 2-sided [-6.324 to 5.548] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; number of participants at 95% CI = 0, 95% CI 2-sided [0.00 to 3.05] — For this particular parameter we have used number of participants at 95% CI computed from Clopper-Pearson method as no risk difference was found between the Triple ½ (GMRx2) vs placebo

18. Other Pre Specified Outcome: Percentage of Participants With eGFR Drop of Over 30% From Randomization to Week 4
Description: The secondary safety outcome is percentage of participants with eGFR drop of over 30% from randomization to Week 4
Time Frame: Randomization to Week 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 0 | 0 | 1
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = -1.59, 95% CI 2-sided [-9.684 to 2.778] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = -1.59, 95% CI 2-sided [-9.684 to 2.590] — 95% confidence intervals for risk difference utilized Newcombe estimation method

19. Other Pre Specified Outcome: Percentage of Participants With Serum Sodium <135mmol/l or >145 mmol/l, and/or Serum Potassium <3.5 mmol/l or >5.5mmol/l at Week 4
Description: The secondary safety outcome is percentage of participants with serum sodium <135mmol/l or >145 mmol/l, and/or serum potassium <3.5 mmol/l or >5.5mmol/l at Week 4
Time Frame: At Week 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 12 | 12 | 4
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 4.27, 95% CI 2-sided [-6.722 to 12.959] — 95% confidence intervals for risk difference utilized Newcombe estimation method
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 3.73, 95% CI 2-sided [-7.158 to 12.133] — 95% confidence intervals for risk difference utilized Newcombe estimation method

20. Other Pre Specified Outcome: Percentage of Participants With Postural Hypotension at Week 4
Description: The secondary safety outcome percentage of participants with postural hypotension at Week 4
Time Frame: At Week 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 7 | 4 | 3
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = 1.43, 95% CI 2-sided [-8.585 to 8.916]
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; Risk Difference (RD) = -1.40, 95% CI 2-sided [-11.077 to 5.161]

21. Other Pre Specified Outcome: Percentage of Participants With Postural Hypertension at Week 4
Description: The secondary safety outcome is percentage of participants with postural hypertension at Week 4
Time Frame: At Week 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo
Number analyzed (Participants) | 113 | 119 | 63
Participants | 19 | 31 | 13
Statistical Analysis 1: Comparison: Triple ¼ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, GEE procedure; Risk Difference (RD) = -3.82, 95% CI 2-sided [-17.664 to 8.366]
Statistical Analysis 2: Comparison: Triple ½ (GMRx2) vs Placebo; Test type: Superiority; p < 0.0001, GEE procedure; LS Means = 5.42, 95% CI 2-sided [-9.040 to 17.981]

ADVERSE EVENTS:
Time Frame: 6 weeks (Single-blind placebo run-in period of 2 weeks and double-blind period of 4 weeks)
Description: The Safety Set is defined as all participants who took at least one dose of study treatment, including during period 1 single-blind placebo run-in
Groups:
- Not Randomized: Participants who were run-in failure and were not randomized
Arm/Group | Triple ¼ (GMRx2) | Triple ½ (GMRx2) | Placebo | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/119 | 0/63 | 0/460
Serious Adverse Events (participants affected / at risk) | 0/113 | 3/119 | 2/63 | 2/460
Other Adverse Events (participants affected / at risk) | 25/113 | 32/119 | 10/63 | 17/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple ¼ (GMRx2) (N=113) | Triple ½ (GMRx2) (N=119) | Placebo (N=63) | Not Randomized (N=460)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple ¼ (GMRx2) (N=113) | Triple ½ (GMRx2) (N=119) | Placebo (N=63) | Not Randomized (N=460)
Blood uric acid increased (Investigations) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 2 (2) | 5 (7) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lipids abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Blood cholesterol decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Low density lipoprotein decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine abnormal (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blood potassium abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
High density lipoprotein abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipids increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT04518306/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04518306/SAP_001.pdf